CLINICAL TRIAL: NCT00654693
Title: A Pilot Study to Evaluate the Performance of Nihon Kohden's NTX Wireless Patient Monitoring System
Brief Title: NTX Wireless Patient Monitoring System
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, James Berry, Professor, Vanderbilt University
Other Study IDs: 080021
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Desaturation; Bradycardia; Tachycardia; Hypertension; Hypotension
Keywords: NTX; Nihon Kohden; mobile monitoring; monitoring; nihon; kohden; monitoring device; remote monitoring; wireless
MeSH Terms: conditions — Bradycardia; Tachycardia; Hypertension; Hypotension | interventions — Hospital Rapid Response Team

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- monitored: patients hospitalized for longer than 24 hours and are located on the 4th, 5th, and 6th floors of the Vanderbilt University Medical Center Round Wing
  Interventions: Other: Rapid Response Team

INTERVENTIONS:
Other: Rapid Response Team — If the subject is experiencing a life threatening change in their vital signs, the Rapid Response Team will be initiated per VUMC protocol.
  Other Names: - attending nurse action per VUMC protocol

SUMMARY:
* Determine the accuracy of the NTX wireless monitoring system alerts
* Evaluate patient compliance with wearing device
* Determine false alarm rates

DETAILED DESCRIPTION:
Approximately 150 patients will have wireless monitors attached to their arm. They will have their vital signs filtered through software that generates alerts and records data. The alert engine will produce pager and application based pop-up alerts which will be sent to the research nurse. Low and high limit alarms will be set according to the published guidelines (Hillman, K. et. Al., Resuscitation 48(2): 105-10, 2001) and adjusted at will by the response team.

During this portion of the study, the following research related procedures will be performed:

* begin continuous vital signs monitoring (BP - 1x per hour, 3 lead ECG -continuous, HR - continuous, SpO2 - continuous)
* PI or Co-PI will review each alert that's generated. The clinical significance will be determined and recorded in the study database
* Record patient's signs and symptoms daily
* Assess concomitant
* Assess AE's, SAEs

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent
* Patients that are hospitalized for longer than 24 hours and are located on the 4th, 5th, or 6th floor of the Vanderbilt University Medical Center Round Wing
* Patients must be ≥18 years of age

Exclusion Criteria:

* ICU patients
* Female subjects who are pregnant
* Patients < 18 years of age
* Patients that have a contradiction for continuous Blood Pressure monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited in the Vanderbilt University Medical Center pre-operative clinic or in the Round Wing, after the effects of anesthesia have worn off. Before performing any trial-related procedures, written Informed Consent and HIPAA authorization will be obtained.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of patient compliance with wearing device | 24 hour minimum post op

SECONDARY OUTCOMES:
Determine accuracy of the NTX wireless monitoring system | duration of patient involvement
Determine false alarm rates | duration of patient involvement

CONTACTS AND LOCATIONS:
Overall Officials: James M Berry, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt University Medical Center Department of Anesthesiology — http://www.vandydreamteam.com